CLINICAL TRIAL: NCT03930524
Title: An Adaptive Preventive Intervention to Optimize the Transition From Universal to Indicated Resources for College Student Alcohol Use
Brief Title: Adaptive Preventive Intervention for College Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Michigan (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006421; R01AA026574 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-04-29 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: College Student Drinking
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Blood Glucose Self-Monitoring; Ethanol; Mass Screening

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Assessment Only (No Intervention): Control
- Early-college Universal (Experimental): Prior to beginning their first semester of college, incoming students will receive personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring surveys over the course of the semester.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM)
- Early-college No Coach (automated email) (Experimental): Students from the early-college universal arm, who flag on one of the self-monitoring surveys are invited to engage in a web-based resource or in-person consultation to improve well-being, with a particular emphasis on alcohol use.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM); Behavioral: Web-BASICS; Behavioral: Health Promotion Consultation
- Early-college Coach (Experimental): Students from the early-college universal arm, who flag on one of the self-monitoring surveys are invited to correspond with an online health coach who will use motivational interviewing strategies to encourage engagement in a web-based resource or in-person consultation to improve wellbeing, with a particular emphasis on alcohol use.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM); Behavioral: Web-BASICS; Behavioral: Health Promotion Consultation; Behavioral: M-Bridge Online Health Coach
- Later-college Universal (Experimental): After beginning their first semester of college, students will receive personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring surveys over the course of the semester.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM)
- Later-college No Coach (automated email) (Experimental): Students from the later-college universal arm, who flag on one of the self-monitoring surveys are invited to engage in a web-based resource or in-person consultation to improve wellbeing, with a particular emphasis on alcohol use.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM); Behavioral: Web-BASICS; Behavioral: Health Promotion Consultation
- Later-college Coach (Experimental): Students from the later-college universal arm, who flag on one of the self-monitoring surveys are invited to correspond with an online health coach who will use motivational interviewing strategies to encourage engagement in a web-based resource or in-person consultation to improve wellbeing, with a particular emphasis on alcohol use.
  Interventions: Behavioral: Personalized Normative Feedback (PNF); Behavioral: Self-Monitoring (SM); Behavioral: Web-BASICS; Behavioral: Health Promotion Consultation; Behavioral: M-Bridge Online Health Coach

INTERVENTIONS:
Behavioral: Personalized Normative Feedback (PNF) — Personalized normative feedback is generated by a process in which: (1) baseline surveys gather respondent information; (2) a computer program links the data with algorithms to select feedback messages; (3) a format for feedback presentation is specified; and (4) the program generates output. Norms will focus on prevalence of drinking, consuming 4/5+ drinks, total number of drinks consumed each week, and maximum drinks consumed. Normative information will be from the national Monitoring the Future (MTF) study college student sample and the University of Minnesota Twin Cities campus. Students will be sent a link to a website where they see their own personal responses in the feedback. Feedback will detail quantity and frequency of drinking (a) reported by the participant him/herself, (b) according to the participant's perception of the descriptive norm for drinking quantity and frequency for the reference group, and (c) reflecting the actual descriptive norm for the reference group.
  Arms: Early-college Coach; Early-college No Coach (automated email); Early-college Universal; Later-college Coach; Later-college No Coach (automated email); Later-college Universal
Behavioral: Self-Monitoring (SM) — Students will be asked to self-report their alcohol use every 2 weeks in response to two main questions (frequency of 4/5+ drinking in the past 2 weeks, frequency of past 2-week 8/10+ drinking), as well as consequences of their drinking. The therapeutic role of SM is two-fold. First, SM facilitates deliberate attention to and reflection on the person's actions, the conditions under which these actions occur, and their consequences (Bandura, 1998; Kanfer, 1970). Hence, SM of drinking behaviors and consequences has the potential to promote awareness of problematic drinking and need for health services. Second, SM affords the opportunity to obtain ongoing information concerning the target behavior, which can be used to inform timely intervention decisions (Nahum-Shani et al., 2016)
  Arms: Early-college Coach; Early-college No Coach (automated email); Early-college Universal; Later-college Coach; Later-college No Coach (automated email); Later-college Universal
Behavioral: Web-BASICS — Web-BASICS is delivered online and responds to individual participant input with the same motivational information and feedback as used in the in-person BASICS intervention. In-person BASICS content (Dimeff et. al., 1999) was developed for online use in studies conducted by Drs. Larimer and Lee (e.g., LaBrie et al., 2013; Lee et al., 2014; Neighbors et al., 2012a). Web-BASICS feedback contains text and graphical feedback regarding students' reported drinking quantity, frequency, peak alcohol consumption, and blood alcohol content (BAC), risks for alcohol problems based on participant family history and consumption patterns, protective behaviors the participant already uses and others he/she might consider, and a tips page with a BAC chart, information on reduced-risk drinking, and where to get more information. Participants can print and/or view their individualized content online for up to 3 months.
  Other Names: Brief Alcohol Screening Intervention for College Students
  Arms: Early-college Coach; Early-college No Coach (automated email); Later-college Coach; Later-college No Coach (automated email)
Behavioral: Health Promotion Consultation — A health promotion consultation via a campus clinic is a confidential exploration of student drug and alcohol use. Health Promotion Consultants help students assess how their alcohol and other substance use affects their life and learn how to make healthier decisions.
  Arms: Early-college Coach; Early-college No Coach (automated email); Later-college Coach; Later-college No Coach (automated email)
Behavioral: M-Bridge Online Health Coach — A health coach will correspond with students via a secure online chat platform, utilizing motivational interviewing strategies to encourage students to consider their values and goals, the possibility of behavior change, and available services. The goal of the dialogue is to motivate the student to access alcohol use interventions (Web-BASICS or an in-person health promotion consultation).
  Other Names: Electronic Bridge to Mental Health Services (eBridge)
  Arms: Early-college Coach; Later-college Coach

SUMMARY:
This research project is designed to promote health among first-year college students by implementing an adaptive sequence of preventive intervention strategies to motivate heavy-drinking college students to access existing resources in order to reduce high-risk alcohol use and negative consequences. If found efficacious, the adaptive preventive intervention (API) has the potential to reduce both the acute negative health consequences (e.g., injury, alcohol poisoning) and long-term health consequences (e.g., alcohol use disorders) of young adult alcohol use, while seeking to leverage technology in order to use campus resources in the most efficient way possible.

DETAILED DESCRIPTION:
College student alcohol use and associated negative consequences are public health problems. In particular, first-year students transitioning to college are at increased risk. Scarce intervention resources must be used as wisely as possible to address these concerns. One way to address heavy drinking while conserving resources is to first utilize universal interventions, identify students at high risk who do not respond well, and then motivate them to engage in indicated intervention. This approach to prevention is 'adaptive' because information about the student in the course of the intervention (e.g., response status) is used to determine whether more resources should be invested to motivate the student to transition to indicated services. The purpose of this project is to implement adaptive preventive intervention (API) that employs cost-effective, technology-based brief interventions to do the following. First, provide a universal personalized normative feedback (PNF) intervention followed by student self-monitoring (SM). Second, motivate students who continue to drink heavily (i.e., 2+ reports of 4/5+ drinks for women/men, or 1 report of 8/10+ drinks for women/men) to transition to additional intervention resources. To optimize the efficacy of this intervention, we will investigate the best timing for delivering the initial universal PNF+SM intervention (i.e., as an inoculation before moving to college vs. once they are experiencing the college context during their first semester). Additionally, we will examine how best to motivate heavy-drinking students to pursue indicated intervention (i.e., via automated emails vs. online interaction with a personal health coach using M-bridge). A sequential multiple assignment randomized trial (SMART) design will be used to address these questions. College students will be randomized to receive PNF either before college begins (2 weeks before classes start) or during the beginning of the first semester (about 3 weeks after they arrive on campus), followed by SM every two weeks during the first semester; these SM assessments will be used to identify heavy-drinking students who remain at risk. Once heavy drinking is identified, the student will be re-randomized to either an automated email or M-bridge health coach to offer indicated intervention resources. The specific aims are to examine: (1) the efficacy of the API compared to an assessment-only control, (2) whether the API can be optimized by altering the timing of the universal intervention and/or the type of message to motivate seeking indicated intervention, and (3) moderators of these effects (e.g., pre-college drinking intentions, high-intensity [compared to binge] drinking during the start of college). Frequency of heavy drinking, alcohol-related consequences, and health services utilization will be assessed prior to the start of classes, and at each follow-up point (the end of the semester, the end of the year, and the following fall). The API to be refined through this project will offer a novel strategy for mitigating both the acute negative health consequences (e.g., injury, alcohol poisoning) and long-term health consequences (e.g., alcohol use disorders) of young adult alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* Incoming college students aged 18-21 at the University of Minnesota will be eligible and randomly selected for participation.

Exclusion Criteria:

* None

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 891 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Patrick, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Labrie JW, Lewis MA, Atkins DC, Neighbors C, Zheng C, Kenney SR, Napper LE, Walter T, Kilmer JR, Hummer JF, Grossbard J, Ghaidarov TM, Desai S, Lee CM, Larimer ME. RCT of web-based personalized normative feedback for college drinking prevention: are typical student norms good enough? J Consult Clin Psychol. 2013 Dec;81(6):1074-86. doi: 10.1037/a0034087. Epub 2013 Aug 12. PMID 23937346
- [Background] Lee CM, Neighbors C, Lewis MA, Kaysen D, Mittmann A, Geisner IM, Atkins DC, Zheng C, Garberson LA, Kilmer JR, Larimer ME. Randomized controlled trial of a Spring Break intervention to reduce high-risk drinking. J Consult Clin Psychol. 2014 Apr;82(2):189-201. doi: 10.1037/a0035743. Epub 2014 Feb 3. PMID 24491072
- [Background] Patrick ME, Boatman JA, Morrell N, Wagner AC, Lyden GR, Nahum-Shani I, King CA, Bonar EE, Lee CM, Larimer ME, Vock DM, Almirall D. A sequential multiple assignment randomized trial (SMART) protocol for empirically developing an adaptive preventive intervention for college student drinking reduction. Contemp Clin Trials. 2020 Sep;96:106089. doi: 10.1016/j.cct.2020.106089. Epub 2020 Jul 25. PMID 32717350
- [Background] Bonar EE, Parks MJ, Gunlicks-Stoessel M, Lyden GR, Mehus CJ, Morrell N, Patrick ME. Binge drinking before and after a COVID-19 campus closure among first-year college students. Addict Behav. 2021 Jul;118:106879. doi: 10.1016/j.addbeh.2021.106879. Epub 2021 Feb 23. PMID 33706071
- [Background] Mehus CJ, Lyden GR, Bonar EE, Gunlicks-Stoessel M, Morrell N, Parks MJ, Wagner AC, Patrick ME. Association between COVID-19-related loneliness or worry and symptoms of anxiety and depression among first-year college students. J Am Coll Health. 2023 Jul;71(5):1332-1337. doi: 10.1080/07448481.2021.1942009. Epub 2021 Jul 9. PMID 34242555
- [Background] Lyden GR, Vock DM, Sur A, Morrell N, Lee CM, Patrick ME. Deeply Tailored Adaptive Interventions to Reduce College Student Drinking: a Real-World Application of Q-Learning for SMART Studies. Prev Sci. 2022 Aug;23(6):1053-1064. doi: 10.1007/s11121-022-01371-7. Epub 2022 May 11. PMID 35543888
- [Background] Carpenter SM, Yap J, Patrick ME, Morrell N, Dziak JJ, Almirall D, Yoon C, Nahum-Shani I. Self-relevant appeals to engage in self-monitoring of alcohol use: A microrandomized trial. Psychol Addict Behav. 2023 May;37(3):434-446. doi: 10.1037/adb0000855. Epub 2022 Jul 14. PMID 35834200
- [Result] Patrick ME, Lyden GR, Morrell N, Mehus CJ, Gunlicks-Stoessel M, Lee CM, King CA, Bonar EE, Nahum-Shani I, Almirall D, Larimer ME, Vock DM. Main outcomes of M-bridge: A sequential multiple assignment randomized trial (SMART) for developing an adaptive preventive intervention for college drinking. J Consult Clin Psychol. 2021 Jul;89(7):601-614. doi: 10.1037/ccp0000663. PMID 34383533

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A random sample of 1500 incoming first-year students were mailed a letter at the end of July 2019 inviting them to participate in the M-bridge study. This was followed by an email invitation sent approximately one week later. Participants enrolled via an online consent form through a link that was provided in the invitations. Study recruitment closed mid-August 2019.
Groups:
- Assessment Only: Assessment Only Control
- Early-college Universal: Prior to beginning first semester of college, incoming students received personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring (SM) surveys over the course of the semester.
  Personalized Normative Feedback: PNF is generated by a process in which: 1) baseline surveys gather respondent information; 2) a computer program links the data with algorithms to select feedback messages; 3) a format for feedback presentation is specified; and 4) the program generates output. Norms focus on prevalence of drinking, consuming 4/5+ drinks, total number of drinks consumed each week, and maximum drinks consumed. Normative information is from the national Monitoring the Future (MTF) study college student sample and the University of Minnesota Twin Cities campus. Students were sent a link to a website where they see their own personal responses in the feedback. Feedback details the quantity and frequency of drinking a) reported by the participant themselves, b) according to the participant's perception of the descriptive norm for drinking quantity and frequency for the reference group, and c) reflecting the actual descriptive norm for the reference group.
  Self Monitoring: Students were asked to self-report their alcohol use every 2 weeks in response to two main questions (frequency of 4/5+ drinking in the past 2 weeks, frequency of past 2-week 8/10+ drinking),as well as consequences of their drinking.
- Early-college No Coach (Automated Email): Students from the early college universal arm, who flagged on one of the self-monitoring surveys were invited to engage in a web-based resource or in-person consultation to improve wellbeing, with a particular emphasis on alcohol use. See PNF and SM described in the early-college Universal arm.
  Web-BASICS is delivered online and responds to individual participant input with the same motivational information and feedback as used in the in-person BASICS intervention. In-person BASICS content (Dimeff et. al., 1999) was developed for online use in studies conducted by Drs. Larimer and Lee (e.g., LaBrie et al., 2013; Lee et al., 2014; Neighbors et al., 2012a). Web-BASICS feedback contains text and graphical feedback regarding students' reported drinking quantity, frequency, peak alcohol consumption, and blood alcohol content (BAC), risks for alcohol problems based on participant family history and consumption patterns, protective behaviors the participant already uses and others he/she might consider, and a tips page with a BAC chart, information on reduced-risk drinking, and where to get more information. Participants can print and/or view their individualized content online for up to 3 months.
  Health promotion consultation via a campus clinic is a confidential exploration of student drug and alcohol use. Health Promotion Consultants help students assess how their alcohol and other substance use affects their life and learn how to make healthier decisions.
- Early-college Coach: Students from the early-college universal arm, who flagged on one of the self monitoring surveys were invited to engage with an online health coach. See PNF and SM described in the early-college universal arm.
  A M-bridge health coach corresponds with students via a secure online chat platform, utilizing motivational interviewing strategies to encourage students to consider their values and goals, possibility of behavior change, and available services. The goal of the dialogue is to motivate students to access alcohol use interventions (Web-BASICS or an in-person health promotion consultation).
  Web-BASICS is delivered online and responds to participant input with the same motivational information and feedback as used in the in-person BASICS intervention. Web-BASICS feedback contains text and graphical feedback regarding students' reported drinking quantity, frequency, peak alcohol consumption, and blood alcohol content (BAC), risks for alcohol problems based on participant family history and consumption patterns, protective behaviors the participant already uses and others they might consider, and a tips page with a BAC chart, information on reduced-risk drinking, and where to get more information.
  Health promotion consultation via a campus clinic is a confidential exploration of student drug and alcohol use. Health Promotion Consultants help students assess how their alcohol and other substance use affects their life and learn how to make healthier decisions.
- Later-college Universal: After beginning their first semester of college, students received personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring surveys over the course of the semester.
  Personalized Normative Feedback: PNF is generated by a process in which: 1) baseline surveys gather respondent information; 2) a computer program links the data with algorithms to select feedback messages; 3) a format for feedback presentation is specified; and 4) the program generates output. Norms focus on prevalence of drinking, consuming 4/5+ drinks, total number of drinks consumed each week, and maximum drinks consumed. Normative information is from the national Monitoring the Future (MTF) study college student sample and the University of Minnesota Twin Cities campus. Students were sent a link to a website where they see their own personal responses in the feedback. Feedback details the quantity and frequency of drinking a) reported by the participant themselves, b) according to the participant's perception of the descriptive norm for drinking quantity and frequency for the reference group, and c) reflecting the actual descriptive norm for the reference group.
  Self Monitoring: Students were asked to self-report their alcohol use every 2 weeks in response to two main questions (frequency of 4/5+ drinking in the past 2 weeks, frequency of past 2-week 8/10+ drinking), as well as consequences of their drinking.
- Later-college No Coach (Automated Email): Students from the later-college universal arm, who flag on one of the self-monitoring surveys are invited to engage in a web-based resource or in-person consultation to improve wellbeing, with a particular emphasis on alcohol use. See PNF and SM described in the later-college universal arm.
  Web-BASICS is delivered online and responds to individual participant input with the same motivational information and feedback as used in the in-person BASICS intervention. In-person BASICS content (Dimeff et. al., 1999) was developed for online use in studies conducted by Drs. Larimer and Lee (e.g., LaBrie et al., 2013; Lee et al., 2014; Neighbors et al., 2012a). Web-BASICS feedback contains text and graphical feedback regarding students' reported drinking quantity, frequency, peak alcohol consumption, and blood alcohol content (BAC), risks for alcohol problems based on participant family history and consumption patterns, protective behaviors the participant already uses and others he/she might consider, and a tips page with a BAC chart, information on reduced-risk drinking, and where to get more information. Participants can print and/or view their individualized content online for up to 3 months.
  Health promotion consultation via a campus clinic is a confidential exploration of student drug and alcohol use. Health Promotion Consultants help students assess how their alcohol and other substance use affects their life and learn how to make healthier decisions.
- Later-college Coach: Students from the later-college universal arm, who flagged on one of the self-monitoring surveys were to engage with an online health coach. See PNF and SM described in the later-college universal arm.
  A M-bridge health coach corresponds with students via a secure online chat platform, utilizing motivational interviewing strategies to encourage students to consider their values and goals, possibility of behavior change, and available services. The goal of the dialogue is to motivate students to access alcohol use interventions (Web-BASICS or an in-person health promotion consultation).
  Web-BASICS is delivered online and responds to participant input with the same motivational information and feedback as used in the in-person BASICS intervention. Web-BASICS feedback contains text and graphical feedback regarding students' reported drinking quantity, frequency, peak alcohol consumption, and blood alcohol content (BAC), risks for alcohol problems based on participant family history and consumption patterns, protective behaviors the participant already uses and others they might consider, and a tips page with a BAC chart, information on reduced-risk drinking, and where to get more information.
  Health promotion consultation via a campus clinic is a confidential exploration of student drug and alcohol use. Health Promotion Consultants help students assess how their alcohol and other substance use affects their life and learn how to make healthier decisions.
Period: Stage 1
Arm/Group | Assessment Only | Early-college Universal | Early-college No Coach (Automated Email) | Early-college Coach | Later-college Universal | Later-college No Coach (Automated Email) | Later-college Coach
Started | 300 | 295 | 0 | 0 | 296 | 0 | 0
Completed | 274 | 254 | 0 | 0 | 253 | 0 | 0
Not Completed | 26 | 41 | 0 | 0 | 43 | 0 | 0
Period: Stage 2 ("Heavy Drinkers")
Arm/Group | Assessment Only | Early-college Universal | Early-college No Coach (Automated Email) | Early-college Coach | Later-college Universal | Later-college No Coach (Automated Email) | Later-college Coach
Started | 0 | 0 | 38 | 37 | 0 | 40 | 43
Completed | 0 | 0 | 36 | 34 | 0 | 33 | 40
Not Completed | 0 | 0 | 2 | 3 | 0 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Early-college Universal: Prior to beginning first semester of college, incoming students received personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring (SM) surveys over the course of the semester.
- Later-college Universal: After beginning their first semester of college, students received personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring surveys over the course of the semester.
- Total: Total of all reporting groups
Arm/Group | Assessment Only | Early-college Universal | Later-college Universal | Total
Number analyzed (Participants) | 300 | 295 | 296 | 891
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (0.218) | 18.1 (0.281) | 18.1 (0.227) | 18.1 (0.243)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 180 | 192 | 556
  Male | 116 | 115 | 104 | 335
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian Non-Hispanic | 31 | 30 | 30 | 91
  Race/Ethnicity: Black Non-Hispanic | 14 | 9 | 9 | 32
  Race/Ethnicity: Hispanic/Latinx | 10 | 15 | 14 | 39
  Race/Ethnicity: White Non-Hispanic | 233 | 229 | 222 | 684
  Race/Ethnicity: Other | 12 | 12 | 21 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 300 | 295 | 296 | 891

OUTCOME MEASURES:

1. Primary Outcome: Binge Drinking
Description: Respondents are asked about the frequency of consuming 4/5+ drinks within a two-hour period in the past 30 days. Questions are based on NIAAA recommended alcohol questions (https://www.niaaa.nih.gov/research/guidelines-and-resources/recommended-alcohol-questions) and Monitoring the Future survey items (http://www.monitoringthefuture.org/).
Time Frame: 3 months
Population: The data reported is for API vs. Assessment Only because the primary aim of the grant was to examine intervention vs. control group differences. As such, this is how the data was analyzed and reported.
Measure: Mean (Standard Deviation); unit: Number of times
Groups:
- Adaptive Preventive Intervention (API): Participants who were randomized to any one of the four APIs embedded in the SMART.
- Assessment Only: Participants who were randomized to the assessment only control arm.
Arm/Group | Adaptive Preventive Intervention (API) | Assessment Only
Number analyzed (Participants) | 591 | 300
Number of times | 1.034 (1.706) | 1.129 (1.843)

ADVERSE EVENTS:
Time Frame: 13 months.
Groups:
- Assessment Only: Participants randomized to the assessment only control arm.
- Early-college Universal: Prior to beginning first semester of college, incoming students received personalized normative feedback (PNF) comparing their experiences to other college students their age, as well as up to 4 self-monitoring (SM) surveys over the course of the semester.
  Personalized Normative Feedback: PNF is generated by a process in which: 1) baseline surveys gather respondent information; 2) a computer program links the data with algorithms to select feedback messages; 3) a format for feedback presentation is specified; and 4) the program generates output. Norms focus on prevalence of drinking, consuming 4/5+ drinks, total number of drinks consumed each week, and maximum drinks consumed. Normative information is from the national Monitoring the Future (MTF) study college student sample and the University of Minnesota Twin Cities campus. Students were sent a link to a website where they see their own personal responses in the feedback. Feedback details the quantity and frequency of drinking a) reported by the participant themselves, b) according to the participant's perception of the descriptive norm for drinking quantity and frequency for the reference group, and c) reflecting the actual descriptive norm for the reference group.
  Self Monitoring: Students were asked to self-report their alcohol use every 2 weeks in response to two main questions (frequency of 4/5+ drinking in the past 2 weeks, frequency of past 2-week 8/10+ drinking), as well as consequences of their drinking.
Arm/Group | Assessment Only | Early-college Universal | Later-college Universal
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/295 | 0/296
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/295 | 0/296
Other Adverse Events (participants affected / at risk) | 0/300 | 0/295 | 0/296

LIMITATIONS AND CAVEATS:
Limitations of the SMART are specified on page 13 of the "Main Outcomes of M-bridge" manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03930524/Prot_SAP_000.pdf